CLINICAL TRIAL: NCT02050347
Title: Phase I Study of Activated T Lymphocytes Expressing Chimeric Antigen Receptors for Therapy of Relapsed CD19-Positive Malignancies Post-Allogeneic Hematopoietic Stem Cell Transplantation Infused Only After Engraftment (CARPASCIO)
Brief Title: Activated T Lymphocytes Expressing CARs, Relapsed CD19+ Malignancies Post-Allo HSCT(CARPASCIO)
Acronym: CARPASCIO
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other); The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Carlos Ramos, Assistant Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-33133 CARPASCIO; CARPASCIO (Other: Baylor College of Medicine)
Record Dates: First submitted 2014-01-29; First posted 2014-01-30 (Estimated); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Non-Hodgkin's Lymphoma; B-Cell ALL; B-Cell CLL
Keywords: CD19.CAR-CD28zeta; chimeric antigen receptor; hematopoietic stem cell transplant
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Leukemia, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Subgroup A1 (Experimental): Patients with residual or relapsed B-cell ALL and with an HLA-matched related donor will receive CD19.CAR-CD28Z T Cells - dose escalation 1
  Interventions: Genetic: CD19.CAR-CD28Z T Cells - dose escalation 2
- Subgroup B1 (Experimental): Patients with other B-cell malignancies and with an HLA-matched related donor will receive CD19.CAR-CD28Z T Cells - dose escalation 1
  Interventions: Genetic: CD19.CAR-CD28Z T Cells - dose escalation 2
- Subgroup A2 (Experimental): Patients with residual or relapsed B-cell ALL and with an unrelated or HLA-mismatched donor will receive CD19.CAR-CD28Z T Cells - dose escalation 2
  Interventions: Genetic: CD19.CAR-CD28Z T Cells - dose escalation 1
- Subgroup B2 (Experimental): Patients with other B cell malignancies and with an unrelated or HLA-mismatched donor will receive CD19.CAR-CD28Z T Cells - dose escalation 2
  Interventions: Genetic: CD19.CAR-CD28Z T Cells - dose escalation 1

INTERVENTIONS:
Genetic: CD19.CAR-CD28Z T Cells - dose escalation 2 — Patients will receive one of the following dose levels:
  Dose Level 1: 5 ×10^5 cells/kg
  Dose Level 2: 1×10^6 cells/kg
  Dose Level 3: 5×10^6 cells/kg
  Arms: Subgroup A1; Subgroup B1
Genetic: CD19.CAR-CD28Z T Cells - dose escalation 1 — Patients will receive one of the following doses:
  Dose Level one: 1x10^5 cells/kg
  Dose Level 2: 5x10^5 cells/kg
  Dose Level 3: 1x10^6 cells/kg
  Arms: Subgroup A2; Subgroup B2

SUMMARY:
Patients have a type of lymph gland cancer called Non-Hodgkin Lymphoma (NHL), acute lymphocytic leukemia (ALL) or chronic lymphocytic leukemia (CLL) (these diseases will be referred to as "lymphoma" or "leukemia"). The lymphoma or leukemia has come back or has not gone away after treatment (including the best treatment known for these cancers). Because there is no standard treatment for this cancer at this time, subjects are asked to volunteer to be in a gene transfer research study using special immune cells.

The body has different ways of fighting infection and disease. No one way seems perfect for fighting cancers. This research study combines two different ways of fighting disease, antibodies and T cells, hoping that they will work together. Both antibodies and T cells have been used to treat patients with cancers; they have shown promise, but have not been strong enough to cure most patients.

T cells can kill tumor cells but there normally are not enough of them to kill all the tumor cells. Some researchers have taken T cells from a person's blood, grown more of them in the laboratory and then given them back to the person.

The antibody used in this study is called anti-CD19. This antibody sticks to cancer cells because of a substance on the outside of these cells called CD19. CD19 antibodies have been used to treat people with lymphoma and leukemia. For this study, the CD19 antibody has been changed so that instead of floating free in the blood it is now joined to the T cells. When an antibody is joined to a T cell in this way it is called a chimeric receptor. The T lymphocytes will also contain CD28, which stimulates T cells and makes them last longer.

Treatment with CD19/CD28 chimeric receptor-T cells has had activity against lymphoma and leukemia when the cells are made from the patients affected by these diseases. In this study, investigators are going to see if this treatment works even better when they make these cells from a healthy stem cell donor. If investigators are not able to collect blood from the stem cell donor, they will collect blood from the subject to make the CD19/CD28 chimeric receptor-T cells.

These CD19/CD28 chimeric receptor T cells are investigational products not approved by the FDA.

The purpose of this study is to find the biggest dose of chimeric T Cells that is safe, to see how long T cells with this chimeric receptor last, to learn what the side effects are, and to see whether this therapy might help people with lymphoma or leukemia after a stem cell transplantation from a donor.

DETAILED DESCRIPTION:
The subject or his/her donor will give blood to make CD19/CD28 chimeric receptor-T cells in the laboratory. These cells will be grown and frozen. To make the T cells, the donor/subject's blood will be stimulated with growth factors to make the T cells grow. To get the CD19 antibody with CD28 to attach to the surface of the T cell, an antibody gene will be inserted into the T cell. This is done with a virus called a retrovirus that has been made for this study and will carry the antibody gene into the T cell. This virus also helps investigators find the T cells in the blood using a special laboratory test. Subjects will be followed for a total of 15 years to see if there are any long term side effects of gene transfer.

When a subject enrolls on this study, s/he will be assigned a dose of CD19/CD28 chimeric receptor-T cells and should not receive other cancer treatment until 6 weeks after cell infusion.

Several studies suggest that the infused T cells need room to be able to proliferate and accomplish their functions and that this may not happen if there are too many other T cells in circulation. Because of that, if the subject's level of circulating T cells is relatively high, s/hemay receive treatment with cyclophosphamide (Cytoxan) and fludarabine (chemotherapy drugs) before the T cells. If the subject is already receiving chemotherapy, this may not be needed.

The subject will be given an injection of cells into the vein through an IV at the assigned dose. The injection will take up to 10 minutes. The research staff will follow the subject in the clinic after the injection for up to 4 hours. If after a 4-6 week evaluation period after the infusion, the subject seems to be experiencing a benefit (confirmed by radiological studies, physical exam and/or symptoms), s/he may be able to receive up to 5 additional doses of the T cells. These additional infusions would be at least 4-6 weeks apart and at the same dose level received the first time or a lower dose.

There will be medical tests during and after treatment. To learn more about the way the CD19 chimeric receptor-T cells are working and how long they last in the body, extra blood will be drawn.

ELIGIBILITY:
Inclusion Criteria:

PROCUREMENT

* Group A: CD19+ B-ALL undergoing allogeneic HSCT or Group B: CD19+ B cell CLL or NHL undergoing allogeneic HSCT
* Life expectancy of ≥12 weeks.
* Patient has an appropriate donor identified for hematopoietic stem cell transplantation

TREATMENT

* Any patient regardless of sex or age with CD19+ B-ALL undergoing allogeneic HSCT (Group A) OR any patient regardless of sex or age with CD19+ B-CLL or NHL undergoing allogeneic HSCT (Group B)
* Residual disease at the time of transplant (bulky or minimal) or post transplant relapse as evidenced by PCR positivity, specific cytogenetic abnormalities, an abnormal population on flow cytometry or increased blasts on bone marrow biopsy or in the peripheral blood. MRD will be defined as detection in blood or marrow of any of the following:

  * Any leukemia specific marker (such as t(9:22) or t(4:11)) documented in the patient's leukemia cells pre transplant on a post transplant evaluation.
  * An immune globulin rearrangement known to be a disease marker for this patient post transplant.
  * A leukemia specific phenotype post transplant at a level of ≥ 0.01%
  * Mixed donor chimerism (any level)
* Life expectancy ≥ 6 weeks
* Karnofsky/Lansky score ≥ 50%.
* Bilirubin ≤ 2 times the upper limit of normal.
* AST ≤ 3 times the upper limit of normal.
* Estimated GFR > 50 mL/min
* Hgb ≥ 7.0 (can be a transfused value)
* Pulse oximetry of > 90% on room air
* Sexually active patients must be willing to utilize one of the more effective birth control methods during the study and for 6 months after ATL infusion. The male partner should use a condom.
* Available allogeneic activated peripheral blood T cell products with >=15% expression of CD19.CAR-CD28ζ determined by flow cytometry (cell dose is based on total cell numbers and not individual antileukemic cell numbers).
* No other investigational antitumor therapy for one month prior to entry in this study.
* Patients or legal guardians must sign an informed consent.

Exclusion Criteria:

* Severe intercurrent infection.
* Evidence of GVHD > grade II.
* Pregnant or lactating.
* History of hypersensitivity reactions to murine protein-containing products.
* Currently taking corticosteroids (>0.5 mg/kg/day prednisone or equivalent) for therapy of GVHD.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-04; Primary Completion 2019-10 (Actual); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with dose limiting toxicity | 6 weeks
  Toxicity is evaluated using CTCAE, version 4.0. Dose limiting toxicity (DLT) will be defined as any of the following that is NOT (1) pre-existing, or (2) due to infection (to which patients with CLL and NHL are predisposed), or (3) due to underlying malignancy, and that may, after consultation with the FDA when indicated, be considered possibly, probably, or definitely related to the study cellular products:
  * Development of Grade III-IV GVHD or Grade II GVHD unresponsive to front line treatment;
  * Non-hematologic DLT is any grade 3 or grade 4 non-hematologic toxicity, including allergic reactions to T cell infusions.
  * Hematologic DLT is defined as any grade 4 hematologic toxicity, including secondary graft failure (as defined per protocol).
  * Patients with evidence of bone marrow disease (metastases or diffuse infiltration) are not evaluable for hematologic dose limiting toxicity.

SECONDARY OUTCOMES:
Number of patients with tumor response | 8 weeks
  We will summarize tumor response by overall response rates. Tumor burden will be measured before and after T cell therapy.
Frequency of T cell products | Up to 15 years
  The frequency of T cells transduced with the vector (T cells expressing CD19.CAR-CD28z) will be summarized at pre and post-infusion time points. Plots of growth curves will be generated to graphically illustrate patterns of T-cell expansion.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Ramos, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

DOCUMENTS (1):
  • Informed Consent Form (2023-02-08): https://cdn.clinicaltrials.gov/large-docs/47/NCT02050347/ICF_000.pdf